CLINICAL TRIAL: NCT04570878
Title: Subcostal Transverse Abdominis Plane Block for Epigastric Cardiac Pacemaker Operation: a Randomized Controlled Trial
Brief Title: Subcostal Transverse Abdominis Plane Block for Epigastric Cardiac Pacemaker Operation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-2007-074-1142
Record Dates: First submitted 2020-09-24; First posted 2020-09-30 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Congenital Heart Disease
Keywords: pacemaker
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SC TAP (Experimental): Bilateral subcostal transverse abdominis plane block will be performed using 0.25% ropivacaine (0.5mL/kg for each side, MAX 20mL for each side) under ultrasound-guidance at the end of surgery.
  Interventions: Procedure: SC TAP
- Control (Active Comparator): No regional block is provided at the end of surgery.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: SC TAP — Bilateral subcostal transverse abdominis plane block will be performed using 0.25% ropivacaine (0.5mL/kg for each side, MAX 20mL for each side) under ultrasound-guidance at the end of surgery.
  Arms: SC TAP
Procedure: Control — No regional block is provided at the end of surgery.
  Arms: Control

SUMMARY:
This prospective randomized controlled trial aims to examine the effect of subcostal transverse abdominis plane block on the postoperative pain and opioid consumption in patients (12y≤ age) who will undergo epigastric cardiac pacemaker operation.

Patients will be allocated to either the SC TAP(subcostal transverse abdominis plane block) group or the control group (no block). Bilateral subcostal transverse abdominis plane block will be performed using 0.25% ropivacaine (0.5mL/kg for each side, MAX 20mL for each side) under ultrasound-guidance at the end of surgery.

The pain score at 10 min after PACU admin, 1, 6, 24 hours after the surgery, the total opioid consumption at 12, and 24 hours after the surgery, the total dose of additional rescue analgesia (intravenous ketololac or nalbuphine) at 12 and 24 hour after the surgery will be recorded.

DETAILED DESCRIPTION:
This prospective randomized controlled trial aims to examine the effect of subcostal transverse abdominis plane block on the postoperative pain and opioid consumption in patients (12y≤ age) who will undergo epigastric cardiac pacemaker operation.

Patients will be allocated to either the SC TAP(subcostal transverse abdominis plane block) group or the control group (no block). Bilateral subcostal transverse abdominis plane block will be performed using 0.25% ropivacaine (0.5mL/kg for each side, MAX 20mL for each side) under ultrasound-guidance at the end of surgery.

The pain score at 10 min after PACU admin, 1, 6, 24 hours after the surgery, the total opioid consumption at 12, and 24 hours after the surgery, the total dose of additional rescue analgesia (intravenous ketololac, acetaminophen, or fentanil) at 12 and 24 hour after the surgery will be recorded.

ELIGIBILITY:
Inclusion Criteria:

- Patients who will undergo epigastric cardiac pacemaker operation. (12≤ years)

Exclusion Criteria:

* Allergy to opioid
* Allergy to local anesthetics
* Coagulation disorder
* Disease in the central and peripheral nervous system
* Significant renal impairment (Creatinine> 3.0 mg/dl)
* Significant hepatic impairment (aspartate transaminase> 120 unit/L, alanine aminotransferase> 120 unit/L)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-07-09 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Pain score, resting | at 10 minutes after the PACU admin
  Pain score at resting is assessed by Numeric rating scale; A numerical rating scale (NRS) requires the patient to rate their pain on a defined scale. For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable.

SECONDARY OUTCOMES:
Pain score, coughing | at 1hour, 6hours, and 24hours after the end of surgery.
  Pain score at coughing is assessed by Numeric rating scale : A numerical rating scale (NRS) requires the patient to rate their pain on a defined scale. For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable.
total opioid consumption at 12, 24 hours after the end of surgery | at 12hours, 24 hours after the end of surgery
  total opioid consumption at 12, 24 hours after the end of surgery (IV Nalbuphine 1mg = IV Morphine 1mg = IV Fentanyl 10mcg (0.01mg)
Total additional dose of acetaminophen | at 12hours, and 24hours after the end of surgery.
  Total additional dose of acetaminophen (mg)
Total additional dose of ketorolac | at 12hours, and 24hours after the end of surgery.
  Total additional dose of ketorolac (mg)
The incidence of side effects of analgesic medications (percent) | within 24 hours after the end of surgery
  The incidence of side effects of analgesic medications: Nausea, Vomit, Constipation, Pruritus, Dizziness, Dry mouth, Sedation
The incidence of side effects of ropivacaine (percent) | within 1 hour after the end of surgery
  The incidence of side effects of ropivacaine: Arrhythmia, Hypotension, ST change, Dizziness, Convulsion
Hospital stay (days) | within 14 days after the end of surgery
  Postoperative hospital stay (days)

CONTACTS AND LOCATIONS:
Locations (1):
- Jin-Tae Kim, Seoul, South Korea